CLINICAL TRIAL: NCT06660628
Title: Large Segmentation Radiotherapy±Deep Inspiratory Breath Hold for Left Sided Breast Cancer, A Real-World Study
Brief Title: Large Segmentation Radiotherapy ± Deep Inspiration Breath Hold(DIBH) for Left Breast Cancer
Acronym: DLLEB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K6433; 2022-PUMCH-B-116 (Other Grant/Funding Number: Peking Union Medical College Hospital)
Record Dates: First submitted 2024-10-22; First posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-09

CONDITIONS: Breast Cancer
Keywords: breast cancer; heart toxicity; DIBH; dose prediction
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surface guided radiation therapy (SGRT) combined with Deep Inspiration Breath Hold (DIBH) technique (Experimental): Patients with left breast cancer treated with Surface guided radiation therapy (SGRT) combined with Deep Inspiration Breath Hold (DIBH) technique
  Interventions: Radiation: Large Segmentation Radiotherapy; Device: DIBH; Device: Surface guided radiation therapy
- laser alignment combined with free breathing treatment (Active Comparator): Patients with left breast cancer treated with traditional laser alignment with free breathing treatment
  Interventions: Radiation: Large Segmentation Radiotherapy; Device: laser alignment; Behavioral: free breathing

INTERVENTIONS:
Radiation: Large Segmentation Radiotherapy — Large Segmentation Radiotherapy±Deep Inspiratory Breath Hold
Device: DIBH — Deep Inspiration Breath Hold
  Arms: Surface guided radiation therapy (SGRT) combined with Deep Inspiration Breath Hold (DIBH) technique
Device: Surface guided radiation therapy — The technology uses modern 3D camera technology to help track and monitor patient movements during set-up and treatment.
  Arms: Surface guided radiation therapy (SGRT) combined with Deep Inspiration Breath Hold (DIBH) technique
Device: laser alignment — Laser systems for virtual simulation and patient positioning in radiotherapy
  Arms: laser alignment combined with free breathing treatment
Behavioral: free breathing — Patients breathe calmly while radiotherapy instead of holding their breath.
  Arms: laser alignment combined with free breathing treatment

SUMMARY:
The study is a single-center, prospective, non-randomized controlled study. The primary objective is to examine the clinical outcomes of utilizing Deep Inspiration Breath Hold (DIBH) in conjunction with hypo-fractionated radiotherapy for patients diagnosed with left-sided breast cancer with a particular focus on its potential to reduce the incidence of cardiac-related clinical and subclinical events.Participants will revieve large segmentation sadiotherapy ± DIBH for left breast cancer and be followed up to gather their clinical cardiac imformation.

ELIGIBILITY:
Inclusion Criteria:

1. 18-70 years old, female, life expectancy > 5 years
2. ECOG 0, 1, 2 points
3. Pathologically diagnosed with left breast cancer and underwent breast-conserving surgery or modified radical mastectomy
4. The patient will receive radiation therapy to the entire breast or chest wall ± the lymphatic drainage area above and below the clavicle ± the lymphatic drainage area in the axilla.
5. No prior neoadjuvant chemotherapy or breast reconstruction.
6. No active cardiac disease, myocardial infarction, or congestive cardiac failure at baseline.
7. Patients can hold their breath for at least 30 seconds after training
8. Patients who can be followed up and agree to follow the plan.
9. Sign the consent form.

Exclusion Criteria:

1. Lesions were observed on both sides of the breast.
2. Diagnosis could not be confirmed by pathology.
3. Distant metastasis was identified.
4. The patient had undergone neoadjuvant chemotherapy or breast reconstruction surgery.
5. Severe cardiac insufficiency; myocardial infarction or uncorrected unstable cardiac arrhythmia or uncorrected unstable angina within the last 3 months; or pericardial disorders
6. The patient's New York Heart Association (NYHA) cardiac classification is within categories 2-4.
7. A history of chronic lung disease, including conditions that may contribute to ductal dilatation, such as chronic obstructive pulmonary disease (COPD) and interstitial pneumonia.
8. Previous mediastinal radiotherapy.
9. Previous or concurrent second primary malignant tumor (except skin cancer that is not a malignant black pigmented tumor, papillary/follicular carcinoma of the thyroid, carcinoma in situ of the cervix, and contralateral non-invasive breast cancer).
10. Irradiation of the lymphatic drainage area of the internal breast is required.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 348 (Estimated)
Dates: Start 2024-08-21 (Actual); Primary Completion 2029-08-21 (Estimated); Study Completion 2034-08-21 (Estimated)

PRIMARY OUTCOMES:
Incidence of subclinical and clinical cardiac events | through study completion, an average of 1 year
  1. Clinical events: newly emerged cardiac diseases after radiotherapy include acute and delayed pericarditis, pericardial effusion and constrictive pericarditis, coronary artery disease, myocardial infarction, cardiac valve disease and arrhythmia.
  2. Subclinical events: new electrocardiogram (ECG) abnormalities, echocardiographic abnormalities, and abnormal elevations of cardiac enzymes after radiotherapy.

SECONDARY OUTCOMES:
Survival | through study completion, an average of 1 year
  Localized regional control rate ,overall survival and disease-related survival.
Cosmetic results | through study completion, an average of 1 year
  cosmetic evaluation(breast-conserving surgery). Excellent: The treated mammary gland is indistinguishable or only slightly different in size, shape, and texture from the contralateral mammary gland. There may be mild thickening of the breast or skin, or scar tissue, but not enough to change the appearance of the colored gland.
  Good: The treated breast is not mildly asymmetric in size or shape compared to the contralateral breast. Thickening or scar tissue in the breast causes only Fair: The treated breast is significantly different in size and shape from the contralateral breast. Such changes involving 1/4 or less of the treated breast are significantly different in appearance from the contralateral breast. The change involves more than 1/4 of the breast tissue.
  Poor: The treated breast is significantly different in appearance from the contralateral breast. The change involves more than 1/4 of the breast tissue or the treated breast has severe sequelae.
Life quality | through study completion, an average of 1 year
  Assessment of patient quality of life by EORTC QLQ-BR23 , a higher score means worse life quality.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol